CLINICAL TRIAL: NCT07354451
Title: Efficacy of Pelvic Nerve Mobilization in Reducing Symptoms of Primary Dysmenorrhea: A Randomized Controlled Trial
Brief Title: Pelvic Nerve Mobilization for Primary Dysmenorrhea
Acronym: PNM-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Collaborators: Health Education Research Foundation (HERF) (Other)
Responsible Party: Principal Investigator, Raheela Kanwal, Assistant professor, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HERF/Research/REC/No-2020-013
Record Dates: First submitted 2025-12-23; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Primary Dysmenorrhea (PD)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: External Pelvic Nerve Mobilization (Experimental): Participants will receive standardized external neurodynamic mobilization techniques targeting the lumbosacral plexus and pudendal nerve pathways. Sessions will be delivered by trained women's health physiotherapists. Each session will last approximately 30 minutes and will be administered three times per menstrual cycle across three consecutive cycles.
  Interventions: Other: External Pelvic Nerve Mobilization
- Arm 2: Sham Mobilization (Sham Comparator): Participants will receive non-therapeutic light manual contact over the lumbosacral and pelvic regions without neural gliding, joint movement, or tissue mobilization. Session duration and therapist interaction will match the intervention group.
  Interventions: Other: Sham Mobilization

INTERVENTIONS:
Other: External Pelvic Nerve Mobilization — Participants will receive a standardized, protocol-driven external neurodynamic mobilization intervention specifically designed to target the lumbosacral plexus and pudendal nerve pathways. Unlike general pelvic manual therapy or routine neural mobilization techniques typically used in musculoskeletal physiotherapy, this intervention incorporates: A predefined sequence of graded neurodynamic maneuvers developed exclusively for this study, combining individually titrated sliders and tensioners based on the participant's symptom irritability and neurodynamic response. Non-internal, purely external application, ensuring a consistent, reproducible method across participants while avoiding variability associated with internal pelvic techniques used in other women's health studies
  Arms: Arm 1: External Pelvic Nerve Mobilization
Other: Sham Mobilization — Participants will receive non-therapeutic light manual contact over the lumbosacral and pelvic regions without neural gliding, joint movement, or tissue mobilization. Session duration and therapist interaction will match the intervention group.
  Arms: Arm 2: Sham Mobilization

SUMMARY:
Primary dysmenorrhea is a highly prevalent condition among young women and is associated with significant pain, reduced quality of life, and academic absenteeism. Although non-steroidal anti-inflammatory drugs are commonly used, many women seek non-pharmacological alternatives due to limited effectiveness or adverse effects. Emerging evidence suggests that altered pelvic neurodynamics may contribute to dysmenorrheic pain.

This randomized controlled trial aims to evaluate the effectiveness of external pelvic nerve mobilization in reducing menstrual pain and associated symptoms among university women with primary dysmenorrhea. Participants aged 18-30 years will be randomly allocated to receive either external pelvic nerve mobilization or a sham manual therapy intervention across three consecutive menstrual cycles. Outcomes will include pain intensity, menstrual distress, quality of life, pelvic tenderness, analgesic consumption, and academic absenteeism.

DETAILED DESCRIPTION:
Primary dysmenorrhea is characterized by painful menstruation in the absence of identifiable pelvic pathology and affects a large proportion of young women. Pain is largely mediated by excessive prostaglandin release, uterine ischemia, and sensitization of pelvic neural pathways. Recurrent nociceptive input may lead to peripheral and central sensitization, exacerbating pain severity.

External pelvic nerve mobilization is a physiotherapy-based neurodynamic intervention designed to restore physiological mobility of pelvic and lumbosacral nerves, reduce neural mechanosensitivity, and modulate nociceptive signaling. Unlike internal pelvic techniques, this approach is entirely external, non-invasive, and suitable for young and student populations.

This single-blind, parallel-group randomized controlled trial will assess whether external pelvic nerve mobilization provides superior pain reduction and functional improvement compared with a sham intervention over three menstrual cycles.

ELIGIBILITY:
Inclusion Criteria:

* Female university students aged 18-30 years
* Regular menstrual cycles (24-35 days)
* Clinically diagnosed primary dysmenorrhea
* Average menstrual pain intensity ≥ 5 on Visual Analog Scale
* Willingness to participate and provide informed consent

Exclusion Criteria:

* Secondary dysmenorrhea (e.g., endometriosis, fibroids, pelvic inflammatory disease)
* History of pelvic or spinal surgery
* Neurological disorders
* Current pregnancy or lactation
* Current physiotherapy or manual therapy treatment
* Contraindications to manual therapy

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Menstrual pain intensity | During the first three days of menstruation at baseline and during the first three days of each menstrual cycle for three consecutive cycles (each cycle = 28 days).
  Menstrual pain intensity will be assessed using a 10-cm Visual Analog Scale (VAS). Participants will rate their average menstrual pain on a scale ranging from 0 to 10, where 0 = no pain and 10 = worst imaginable pain. Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
Analgesic consumption | Baseline (Cycle 0; prior menstrual cycle, defined as 28 days) and during menstruation for Cycles 1, 2, and 3 (each cycle = 28 days).
  Analgesic consumption will be measured as the total number of analgesic doses consumed for menstrual pain management. Participants will record the type and number of doses taken during menstruation. Higher values indicate greater medication use.
Academic absenteeism | Baseline (Cycle 0; prior menstrual cycle, defined as 28 days) and during menstruation for Cycles 1, 2, and 3 (each cycle = 28 days).
  Academic absenteeism will be assessed as the total number of hours missed from academic activities due to menstrual pain, as self-reported by participants. Higher values indicate greater absenteeism.
DAILY RECORD OF SEVERITY OF PROBLEMS | Baseline (Cycle 0; daily for a full 28-day menstrual cycle) and daily across Cycles 1, 2, and 3 (each cycle = 28 days).
  Menstrual-related symptoms will be assessed using the Daily Record of Severity of Problems (DRSP) questionnaire. The DRSP evaluates physical, emotional, and behavioral symptoms on a 6-point Likert scale (1 = not at all to 6 = extreme), with higher scores indicating greater symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- International Institute of Science Arts and Technology, Sialkot, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains sensitive participant information, and there is a risk of re-identification. The study does not include a data-sharing plan or a secure mechanism for providing external access.